CLINICAL TRIAL: NCT05648331
Title: Wheelchair Use in Patients With Lower Limb Amputation
Brief Title: Wheelchair Use in Patients With Amputation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Gaziler Physical Medicine and Rehabilitation Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Yasin Demir, Associated Proffessor, Gaziler Physical Medicine and Rehabilitation Education and Research Hospital
Other Study IDs: 30
Record Dates: First submitted 2022-12-05; First posted 2022-12-13 (Actual); Last update posted 2023-01-03 (Actual); Status verified 2022-12

CONDITIONS: Amputation, Wheelchair

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
There are no specific criteria for wheelchair use in patients with lower extremity amputations. The main purpose of this study is to determine the characteristics of wheelchair use in lower extremity amputee patients. In addition, it is aimed to determine the reasons for using and not using a wheelchair, and what type of wheelchair is needed.

DETAILED DESCRIPTION:
There are no specific criteria for chair use in patients with lower extremity amputations. The main purpose of this study is to determine the characteristics of wheelchair use in lower extremity amputee patients. In addition, it is aimed to determine the reasons for using and not using a wheelchair, and what type of wheelchair is needed. Thus, it is thought that the main points to be considered while prescribing a wheelchair in patients with amputation can be determined.

Patients with traumatic unilateral or bilateral lower extremity amputation who are hospitalized or applied to outpatient clinics will be included in the study. Demographic and clinical characteristics of the patients will be recorded. Current age, time since the injury (in months), occupation, etiology (mine,rocket launcher, rifle, shrapnel, etc.), amputation level, amputation side, accompanying upper extremity problem, last operation reason, and activity level, knee joint type (hydraulic, simple microprocessor, other microprocessor), foot type (carbon, hydraulic, microprocessor controlled), socket-suspension type, daily use of prosthesis (hour/day), use of assistive device or AFO, how long he/she has been using a wheelchair, the type of wheelchair (light manual, active, battery powered), the reason for using a wheelchair, the reason for not using, the frequency of using a wheelchair, the upper extremity problem/pain while using the chair will be recorded.

ELIGIBILITY:
Inclusion Criteria:

age between 18 and 65 years, time since amputation ≥ 6 months, unilateral or bilateral LLA above the ankle level

Exclusion Criteria:

None

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The age limit of 18-65 years was determined because age may affect the age-related activity level and isokinetic measurements of the patients.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-01-10 (Estimated); Primary Completion 2023-02-28 (Estimated); Study Completion 2023-03-30 (Estimated)

PRIMARY OUTCOMES:
Wheelchair type | through study completion, an average of one and a half months
  Active, light, powered

SECONDARY OUTCOMES:
Reason for wheelchair use | through study completion, an average of one and a half months
  Mobility, upper extremity pain, transfer

CONTACTS AND LOCATIONS:
Locations (1):
- Gaziler Physical and Rehabilitation Medicine Training and Research Hospital, University of Health Sciences, Ankara, Turkey (Türkiye)